CLINICAL TRIAL: NCT03994848
Title: Pulmonary Prehabilitation With Incentive Spirometry in Patients Undergoing One-Lung Ventilation and the Effect on Postoperative Lung Function: A Randomized-Controlled Trial
Brief Title: Incentive Spirometry Prehabilitation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jeffry B. Dobyns, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Spirometry
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Spirometry Group (Experimental)
  Interventions: Behavioral: Spirometry Group

INTERVENTIONS:
Behavioral: Spirometry Group — Patients that are provided the incentive spirometer pre-operatively and instructed to use it for 4 cycles of 10 spirometry attempts on the day prior to surgery
  Arms: Spirometry Group

SUMMARY:
Postoperative pulmonary complications (PPCs) are the most common complication following thoracic surgery. PPCs are associated with prolonged hospital stay, increased morbidity, mortality, ICU admission, and healthcare costs (Azhar, 2015). Current preoperative optimization in this patient group includes smoking cessation and management of Chronic Obstructive Pulmonary Disease with inhaled bronchodilators and inhaled steroids as indicated. There have been studies using preoperative incentive spirometry in patients undergoing laparotomy with conflicting results, but scant data on its use in patients undergoing one-lung ventilation (Tyson, et al., 2015; Cattano, et al., 2010). A study from 2013 investigated the effectiveness of incentive spirometry in patients following thoracotomy and found conflicting results, without significant improvement in lung function or reduction in PPCs, but a larger difference in frequency of PPC was noted, indicating possible benefit to intervention and a need for further study (Agostini, et al., 2013). Volume-based incentive spirometry pre- and postoperatively has also been found to improve pulmonary function and diaphragm excursion in patients undergoing laparoscopic surgery (Alaparthi, et al., 2016).

Patients customarily receive an incentive spirometer for use postoperatively in the PACU. There is scant data in the thoracic surgery population concerning prehabilitation by dispensing the incentive spirometer at the PACT evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thoracic surgery procedures involving one-lung ventilation
* open thoracotomy
* Video-assisted thoracoscopic surgery (VATS)
* Robotic-assisted thoracoscopic surgery (RATS)
* Procedures to include: Lung resection for any purpose, esophagectomy, thymectomy
* Patients undergoing esophagectomy performed by a general surgeon
* Patients willing and able to independently perform incentive spirometry

Exclusion Criteria:

* Trauma patients
* Lung Volume reduction surgery (LVRS)
* In-Patients
* Patients not undergoing one-lung ventilation
* Patients undergoing thoracoabdominal aortic aneurysm repair
* Transhiatal esophagectomy (does not involve one-lung ventilation)
* Lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Lung Volumes | From the time of admission to the pre-operative holding area to 72 hours post-operatively
  Mean Lung Volumes

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Dobyns, DO, MSHA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No